CLINICAL TRIAL: NCT04381572
Title: The Impact of High Fidelity Simulation on Stress Level in Medical Students.
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Piotr Palaczyński, Principal Investigator, Medical University of Silesia
Other Study IDs: SSS-01
Record Dates: First submitted 2020-05-02; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Stress, Physiological; High Fidelity Simulation Training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High fidelity simulation training: Group consisting of medical students scheduled to undergo high fidelity medical simulation as a part of standard scholastic program.
  Interventions: Behavioral: High fidelity simulation training

INTERVENTIONS:
Behavioral: High fidelity simulation training — At the beginning of scheduled classes in the simulation center, students were placed sitting at rest for 30 min. In each team a leader was chosen. Other team members were also assigned detailed functions. Before starting the scenario, participants were oriented for 10 -15 minutes by a physician instructor about the simulation room setup and manikin features. The simulated scenarios were performed using a high fidelity computer-based manikin simulator, with the possibility of remote control of vital signs. All medications and equipment required during the clinical scenarios were available. The scenario used was prepared and validated by experienced simulation instructors. All student groups were given the same standardized scenario.

SUMMARY:
High fidelity simulation (HFS) is an established method of training in various fields of medicine, especially emergency medicine, anesthesiology and intensive therapy. One of the benefits of HFS as an educational tool is the protective environment, where the risk of error do not bring harm to the patients.

It is proven that HFS is successful in acquisition of new knowledge and skills and may facilitate positive behavioral change in medical students. However, this education method may cause elevated stress levels as well as other physiological reactions. Other than sympathetic nervous system reactions such as heart rate and blood pressure, there are a few laboratory stress level markers such as cortisol, alpha-amylase, testosterone and secretory immunoglobulin A. Our aim was to evaluate the change of stress level induced by high-fidelity simulation in medical students.

ELIGIBILITY:
Inclusion Criteria:

* willingness to take part in the study

Exclusion Criteria:

* pregnancy,
* active infections
* diseases of immune system
* metabolic or endocrine disturbances
* current use of any medication (except for oral contraceptives)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical faculty students (fifth and sixth year) scheduled to undergo high fidelity medical simulation as a part of standard scholastic program.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Α-amylase activity in saliva [U/ml] | 120 minutes
  Saliva was collected using a disposable Salivette tube (Sarstedt AG & Co, Germany) by placing a sterile tampon under the tongue or chewing for 30-45 seconds. Next the tube was centrifuged (1000 x g for 10 min.) to obtain a ready to test saliva supernatant. Samples were frozen after centrifugation at - 85°C until performing laboratory tests. Α-amylase activity assay was performed by a static method with AMYLAZA kit (Aqua-Med Łodz, Poland). The samples were diluted 100 times using 0,9% chloride solution. 2-chloro-4-nitrofenylo-maltotrioside is a substrate in this method. The reaction was performed in pH 6,0 MES buffer at 37 ° C rendering a colored reaction product. The product was then analyzed via spectrophotometry at 405 nm.
Secretory immunoglobulin class A concentration in saliva [ug/ml] | 120 minutes
  Saliva was collected using a disposable Salivette tube (Sarstedt AG & Co, Germany) by placing a sterile tampon under the tongue or chewing for 30-45 seconds. Next the tube was centrifuged (1000 x g for 10 min.) to obtain a ready to test saliva supernatant. Samples were frozen after centrifugation at - 85°C until performing laboratory tests. Determination of secretory immunoglobulin class A (sIgA) concentration was established using an ELISA (Immunodiagnostic AG, Germany). The analytical procedure was carried out in accordance to the instructions provided by the manufacturer in the user manual. Absorbance readings were taken using a μQuant reader (BioTek, USA), the results were processed using the KCJunior program (BioTek, USA).
Cortisol concentration in saliva [ng/ml] | 120 minutes
  Saliva was collected using a disposable Salivette tube (Sarstedt AG & Co, Germany) by placing a sterile tampon under the tongue or chewing for 30-45 seconds. Next the tube was centrifuged (1000 x g for 10 min.) to obtain a ready to test saliva supernatant. Samples were frozen after centrifugation at - 85°C until performing laboratory tests.
  The commercial ELISA (Diapra, Italy) were used to determine the concentration of cortisol in saliva. The analytical procedure was carried out with accordance to the manufacturer's instructions in the technical manual supplied with the kit. Absorbance readings were taken using a μQuant reader (Biotek, USA), while results were processed using KCJunior (Biotek, USA).
Testosterone concentration in saliva [pg/ml] | 120 minutes
  Saliva was collected using a disposable Salivette tube (Sarstedt AG & Co, Germany) by placing a sterile tampon under the tongue or chewing for 30-45 seconds. Next the tube was centrifuged (1000 x g for 10 min.) to obtain a ready to test saliva supernatant. Samples were frozen after centrifugation at - 85°C until performing laboratory tests.
  The commercial ELISA (Diapra, Italy) was used to determine the concentration of testosterone in saliva. The analytical procedure was carried out with accordance to the manufacturer's instructions in the technical manual supplied with the kit. Absorbance readings were taken using a μQuant reader (Biotek, USA), while results were processed using KCJunior (Biotek, USA).
Total protein concentration [mg/ml] | 120 minutes
  Saliva was collected using a disposable Salivette tube (Sarstedt AG & Co, Germany) by placing a sterile tampon under the tongue or chewing for 30-45 seconds. Next the tube was centrifuged (1000 x g for 10 min.) to obtain a ready to test saliva supernatant. Samples were frozen after centrifugation at - 85°C until performing laboratory tests. To determine the total protein concentration the Lowry method was used. This method base on the reactions between peptide bonds, tyrosine and Folin-Ciocalteu reagent. The absorbance of the resulting color was read at a wavelength of 650-750 nm, 30 minutes after the addition of the reagent. Bovine serum albumin water solution (BSA - Sigma Aldrich, Germany) at slightly basic pH was used as standard.

SECONDARY OUTCOMES:
Heart rate [bpm] | 120 minutes
  Heart rate was measured using a cardiomonitor (Infinity Delta, Dräger; Germany).
Blood pressure [mmHg] | 120 minutes
  Blood pressure was measured using a cardiomonitor (Infinity Delta, Dräger; Germany).
Saturation [%] | 120 minutes
  Saturation level was measured using a cardiomonitor (Infinity Delta, Dräger; Germany).

CONTACTS AND LOCATIONS:
Locations (1):
- Samodzielny Publiczny Szpital Kliniczny nr 1, Zabrze, Silesian Voivodeship, Poland